CLINICAL TRIAL: NCT06482905
Title: A Phase I, Open-Label, Single/Multiple Dose, Dose-escalation Study to Evaluate the Safety, Tolerability and Antitumor Activity of TX103 CAR-T Cell Injection (TX103) in Subjects With Recurrent or Progressive Grade 4 Glioma.
Brief Title: Safety and Efficacy Study of TX103 CAR-T Cell Therapy for Recurrent or Progressive Grade 4 Glioma.
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Tcelltech Inc. (Industry)
Collaborators: Beijing Tiantan Hospital (Other); Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TX103T-RG008
Record Dates: First submitted 2024-06-15; First posted 2024-07-01 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-04

CONDITIONS: High-grade Glioma; WHO Grade Ⅳ Glioma
MeSH Terms: conditions — Glioma | interventions — Immunotherapy, Adoptive; Injections

STUDY DESIGN:
Intervention Model Description: a "3+3" design is used to determine Maximum Tolerated Dose (MTD) and the recommended phase 2 dose (RP2D)
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Safety Run-In (Experimental): Single-dose administration of TX103 via intraventricular(ICV) or intracavitary (ICT) .
  Interventions: Biological: Anti-B7-H3 Chimeric Antigen Receptor T-Cell (CAR-T Cell) Injection/TX103
- Cohort A Single delivery route(Multi-dose) (Experimental): Administration of TX103 via intraventricular(ICV) on Days 1 and 8 in a 21-day treatment cycle.
  Interventions: Biological: Anti-B7-H3 Chimeric Antigen Receptor T-Cell (CAR-T Cell) Injection/TX103
- Cohort B Dual delivery route(Multi-dose) (Experimental): Administration of TX103 on Day 1 via intracavitary (ICT) and on Day 8 via intraventricular(ICV) in a 21-day treatment cycle.
  Interventions: Biological: Anti-B7-H3 Chimeric Antigen Receptor T-Cell (CAR-T Cell) Injection/TX103

INTERVENTIONS:
Biological: Anti-B7-H3 Chimeric Antigen Receptor T-Cell (CAR-T Cell) Injection/TX103 — Safety Run-In: Dose:6×10^7 CAR+ T cells
  Cohort A Single delivery route(Multi-dose)、Cohort B Dual delivery route(Multi-dose)： 3+3 dose escalation design： Dose Level 1: 6×10^7 CAR+ T cells Dose Level 2: 1.5×10^8 CAR+ T cells Dose Level 3: 2.5×10^8 CAR+ T cells

SUMMARY:
This is a phase I, open-Label, single/multiple dose, dose-escalation study to evaluate the safety, tolerability and antitumor activity of anti-B7-H3 CAR-T cell injection (TX103) in subjects with recurrent or progressive Grade 4 Glioma.The study also plan to explore the Maximum Tolerated Dose (MTD) and determine the Recommended Phase II Dose (RP2D) of the CAR-T cell therapy.

DETAILED DESCRIPTION:
Eligible subjects will be enrolled into two sequential dose-escalating cohorts (i.e., A and B), and will be administrated TX103. Cohort A will receive TX103 exclusively through intraventricular (ICV) delivery, while cohort B will undergo dual intracavitary (ICT) and ICV delivery. Patients in each individual cohort will receive two TX103 infusions on Day 1 and 8 respectively, followed by a 14-day observation period in a 21-day treatment cycle.

Three escalating dosage levels are planned for each cohort. Both Cohorts A and B will adopt the traditional 3+3 dose escalation design with each dose level enrolled with 3 to 6 patients. The starting dose will be 6 × 10^7 CAR+ T cells (i.e., Dose Level 1, DL1). Dose limiting toxicities (DLTs) will be assessed during the first cycle .

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must voluntarily participate in the study and sign a written informed consent document; subjects should be willing and able to follow and complete study procedures.
2. Male or female subjects aged 18 to 75 years (both inclusive).
3. Subject must have histologically diagnosed grade 4 glioma, such as glioblastoma, grade 4 astrocytoma, diffuse hemispheric glioma, according to 2021 WHO Classification of Tumors of the CNS. Subjects must have had experienced disease recurrence or progression* after surgery combined with Stupp regimen (concurrent radiotherapy and temozolomide (TMZ) followed by adjuvant TMZ) and are not candidate for re-resection. For subjects harboring specific gene mutations, such as NTRK gene fusion or BRAF V600E mutation, they must have also progressed on corresponding mutation-directed therapies before enrollment.

   * Disease recurrence or progression must be confirmed by radiographic or histopathological diagnosis.
4. Subjects with confirmed B7-H3 positive* (≥30%) tumor expression by immunohistochemistry (IHC) in either primary or recurrent tumor tissue.

   *B7-H3 positive rate is defined as the percentage of B7-H3 positive tumor cells in non-necrotic tumor tissue.
5. Subjects with KPS score of ≥60.
6. Subjects should have adequate venous access for collection of peripheral blood mononuclear cells (PBMCs).
7. Subjects with left ventricular ejection fraction (LVEF) ≥ 40% within one month prior to the first dose.
8. Subjects with oxygen saturation ≥95% under the resting state.
9. Subjects with adequate organ function, as indicated by laboratory test results that meet the following criteria:

   * Hematological function: Absolute neutrophil count (ANC) ≥1.5×109/L, hemoglobin (Hb) ≥90g/L, platelet count (PLT) ≥100×109/L, absolute lymphocytes count (ALC) ≥0.15×109/L. Blood transfusion, granulocyte (macrophage) colony stimulating factor, recombinant human erythropoietin, recombinant human thrombopoietin, platelet receptor agonist, recombinant human interleukin-11, and other supportive treatments are prohibited within 14 days before the test.
   * Liver function: Total bilirubin (TBIL) ≤ 1.5 × ULN, patients with Gilbert's syndrome (persistent or recurrent hyperbilirubinemia, presenting as unconjugated bilirubin in the absence of evidence of hemolysis or liver pathology) Except for elevated erythrocytes; alanine aminotransferases (ALT) and aspartate aminotransferase (AST) ≤2.5×ULN.
   * Renal function: serum creatinine (Scr) ≤1.5×ULN.
   * Coagulation function (in the absence of anticoagulant therapy): prothrombin time (PT) or activated partial thromboplastin time (APTT) or international normalized ratio (INR) ≤ 1.5×ULN.
   * Female subjects of childbearing potential must have a negative serum pregnancy test at screening and if a positive urine test or a negative result cannot be confirmed by urine test.
10. Women of childbearing potential (which refer to women who have not been surgically sterilized and pre-menopausal women) should use highly effective and reliable method of contraception (refer to Section 5.3 for contraception method) from the start of the study until 6 months after the last dose of the study drug; sexually active male subjects, if no vas deferens for ligation, consent must be given to the use of highly effective and reliable method of contraception from the start of the study until 6 months after the last dose of the study drug.

Exclusion Criteria:

1. Pregnant or breastfeeding female subjects.
2. Subjects with viral infection during the screening period:

   * Serum HIV antibody positive, treponema pallidum serology positive; OR
   * Hepatitis B surface antigen (HBsAg) positive and peripheral blood HBV DNA test value exceeds the normal range; OR
   * Hepatitis C virus (HCV) antibody positive and peripheral blood HCV RNA positive.
3. Medical history and concomitant diseases:

   * Subjects who have received carmustine extended-release implantation surgery within 6 months;
   * Subjects with known or suspected active autoimmune diseases, including but not limited to Crohn's disease, rheumatoid arthritis, systemic lupus erythematosus, etc.;
   * Subjects who are receiving systemic immunosuppressive agents or subjects who need to use immunosuppressive agents for a long-time during treatment, except for intermittent topical, inhaled, or intranasal glucocorticoid therapy;
   * Subjects with uncontrolled mental disorders, or who, in the Investigator's opinion, have a medical history or a history of mental states that may increase the risks associated with study participation or study drug administration, or that may interfere with the results;
   * The toxicity and side effects caused by previous treatment have not recovered to ≤ grade 1 (per CTCAE 5.0); except for alopecia and other tolerable events judged by the Investigator;
   * Subjects who have participated in other interventional clinical studies within the past 1 month;
   * Subjects who have previously received CAR-T cell therapy or other gene therapy*;
   * Subjects with any serious or poorly controlled disease that, in the opinion of the Investigator, may increase the risk associated with study participation, study drug administration, or affect the subject's ability to receive study drug, including but not limited to cardiovascular and cerebrovascular diseases, renal insufficiency, pulmonary embolism, coagulopathy or requiring long-term anticoagulant therapy, active infection or uncontrollable infection requiring long-term systemic treatment;
   * Subjects with other malignant tumors in the past 3 years or at present, except for non-melanoma skin cancer, carcinoma in situ (such as cervix, bladder and breast cancer).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2024-09-04 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Safety：Incidence of Dose Limiting Toxicity (DLT) | 28 days after the first TX103 infusion.
  Type, incidence, and severity of dose limiting toxicities (DLTs) within 28 days after the first TX103 infusion.
Safety：Incidence and severity of adverse events (AEs) | six months post CAR-T cells infusion.
  To evaluate the possible adverse events after TX103 infusion, including the incidence, and severity of AEs.

SECONDARY OUTCOMES:
Overall survival (OS) | 6 and 12 months post CAR-T cells infusion.
  The proportion of subjects who have survived for more than 6 and12 months since the diagnosis of recurrent or progressive Grade 4 Glioma.
Post-relapse survival (PRS) | 6 and 12 months post CAR-T cells infusion.
  The proportion of subjects who have survived for more than 6 and12 months since the diagnosis of recurrent or progressive Grade 4 Glioma.
Progression Free Survival (PFS) | 1 year post CAR-T cells infusion.
  To evaluate the time from the start of TX103 therapy to disease progression (according to RANO2.0 criteria) or death from any cause, whichever occurs first. The proportion of progression-free subjects from the beginning of TX103 therapy to a fixed time point (6 months) after treatment (6-Mon PFS) will also be evaluated.
Disease Control Rate (DCR) | 1 year post CAR-T cells infusion.
  To evaluate the proportion of subjects who achieved CR/PR/SD in the best overall response according to RANO2.0 criteria.
Duration of disease control (DDC) | 1 year post CAR-T cells infusion.
  To evaluate the time from the first evaluation of tumor as CR, PR or SD to the first evaluation of PD or death from any cause.
Objective response rate (ORR) | 1 year post CAR-T cells infusion.
  To evaluate the proportion of subjects who achieved CR/PR in the best response condition according to RANO2.0 criteria.
Time to Remission (TTR) | 1 year post CAR-T cells infusion.
  To evaluate the time from the start of treatment to the first remission (CR/PR).
Duration of Response (DOR) | 1 year post CAR-T cells infusion.
  DOR after TX103 infusion, defined as the time from the first evaluation of the tumor as CR or PR to the first evaluation of PD or death from any cause.
Neurological function evaluated by NANO scale | 1 year post CAR-T cells infusion.
  Change in neurological function from baseline.
Quality of life score | 1 year post CAR-T cells infusion.
  Change in Quality of life score from baseline.

OTHER OUTCOMES:
The immunogenicity of TX103 | up to 12 months.
  Drug antibody (ADA) positive rate after infusion of TX103 cells.
The positive rate of replication competent lentivirus tests | up to 15 years.
  Detect replication competent lentivirus (RCL).
Incidence of Secondary Malignancies | up to 15 years.
  The frequency and occurrence of new, distinct cancerous growths that develop as a result of TX103.
Peak Concentration (Cmax) of TX103 CAR gene | Up to 12 months.
  Peak Concentration (Cmax) of TX103 CAR gene
Area under the concentration versus time curve (AUC) of TX103 CAR-T cells | Up to 12 months.
  Area under the concentration versus time curve (AUC) of TX103 CAR-T cells
Peak concentration of cytokines | Up to 12 months.
  Peak concentration of IL-2, IL-4，IL-6, IL-8，IL-10，IFN-γ， TNF-a

CONTACTS AND LOCATIONS:
Overall Officials: Gangxiong Huang, MD, Study Director — Tcelltech Inc.
Locations (4):
- United States (3):
  - Mayo Clinic in Arizona, Phoenix, Arizona
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Mayo Clinic in Rochester, Rochester, Minnesota
- Beijing Tiantan Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No